CLINICAL TRIAL: NCT04326530
Title: Use of a Modern Breath Sampling System (the Pneumopipe® Combined With an Array of E-nose Sensors) for the Prediction of Treatment Response in Persistent Asthmatic Children
Acronym: Pneumo-Pred
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Istituto per la Ricerca e l'Innovazione Biomedica (Other)
Collaborators: Campus Bio-Medico University (Other)
Responsible Party: Principal Investigator, Stefania La Grutta, MD, Senior Researcher, Istituto per la Ricerca e l'Innovazione Biomedica
Other Study IDs: 3/2020
Record Dates: First submitted 2020-03-26; First posted 2020-03-30 (Actual); Last update posted 2022-12-19 (Actual); Status verified 2022-12

CONDITIONS: Asthma in Children

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Persistent asthmatic children: 150 steroid-naive, persistent asthmatic children enrolled during their first consultation at the IRIB-CNR outpatient clinic.
  They will underwent three visits:
  1. screening visit (-2 days);
  2. baseline visit (day 0);
  3. last visit (+90 days).
  They will be treated with controller medications according to GINA recommendations (http://ginasthma.org).
  Interventions: Device: Pneumopipe® (European patent 12425057.2, Rome, Italy); Other: Other assessments

INTERVENTIONS:
Device: Pneumopipe® (European patent 12425057.2, Rome, Italy) — Collection of VOCs on a cartridge after that the child has normally breathed in it for 3 min, both at the baseline and at the last visit.
Other: Other assessments — * Spirometry, both at the baseline and at the last visit.
  * 24-hour urine collection, both at the baseline and at the last visit.

SUMMARY:
Due to a large disease heterogeneity, the proper management of childhood asthma may be a challenging task. Despite the screening of lung function is a fundamental tool, spirometry alone may not allow a reliable prediction of the disease prognosis, such as treatment response and asthma exacerbations.

Recently, it has been shown that the detection of volatile organic compounds (VOCs) in exhaled breath (Breathomics) is able to predict asthma exacerbations and to discriminate children with persistently controlled asthma from those with uncontrolled asthma. These studies have been realized through gas chromatography / mass spectroscopy techniques, which also provide information on specific compounds useful for pathophysiologic research; however, they are expensive and time consuming.

An alternative approach, scarcely adopted so far, is based on cross-reactive nonspecific sensor arrays (e-noses), which may provide valuable information on disease status through pattern recognition algorithms or discriminant analyses of the global sensor response pattern (breath-fingerprint). In particular, the Pneumopipe® (European patent 12425057.2, Rome, Italy) is a recent and innovative device allowing direct absorption of VOCs on a cartridge after an individual has normally breathed in it for 3 min. It is a very simple and cheap procedure, suitable for non-collaborative populations. Moreover, cartridges may be preferable over sampling bags in terms of preservation and transportability. This modern breath sampling system provides repeatable measurements, and negligible overlap has been observed with information provided by spirometry.

The main objective of the present study is to assess whether baseline (pre-treatment) spirometry and e-nose measurements may predict asthma prognosis in persistent asthmatic children, in terms of response to the prescribed treatment with inhaled steroid (ICS), and to provide simple rules for discriminating treatment responders and non-responders. The secondary aim is to assess e-nose ability to predict asthma exacerbations, disease control and adherence.

ELIGIBILITY:
Inclusion criteria:

* male or female gender
* age between 6 and 16 years
* first asthma diagnosis according to GINA recommendations (http://ginasthma.org), including assessment of the history of respiratory symptoms (wheezing, shortness of breath, chest tightness and cough) and environmental exposures (smoke, mold, vehicular traffic), spirometry (FEV1/FVC<0.90 at baseline, >12% FEV1 increase from baseline after bronchodilator inhalation) and skin prick tests.

Exclusion criteria:

* exacerbations requiring oral corticosteroids in the last four weeks
* use of controller medications (leukotriene receptor antagonists and/or inhaled corticosteroids) in the last four weeks
* respiratory infections in the last four weeks
* immunological, metabolic, cardiac or neurological diseases
* major malformations of the respiratory system
* active smoking.

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 150 steroid-naive, persistent asthmatic children enrolled during their first consultation at the IRIB-CNR outpatient clinic.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Treatment decision at the last visit | 90 days
  ICS dose step-down (type-1 mismatching, i.e. unexpectedly good prognosis), same ICS dose (perfect matching, i.e. expected prognosis) or ICS dose step-up (type-2 mismatching, i.e. unexpectedly bad prognosis).

SECONDARY OUTCOMES:
Asthma exacerbations | 90 days
  Occurrence of asthma exacerbations in the time interval between the baseline and the last visit.
CACT-ACT | 90 days
  Childhood Asthma Control Test (C-ACT, for children aged 6-11) or Asthma Control Test (ACT, for children aged 12-16). The total score ranges from 0 (poor asthma control) to 27 (optimal asthma control).
Treatment adherence | Day 0; 90 days
  Change in urinary cortisol levels (last vs baseline visit);
Treatment adherence | 90 days
  9-item Medication Adherence Rating Scale (MARS-9). The total score ranges from 5 to 45. Higher scores indicate higher self-reported adherence.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fasola S, Ferrante G, Sabatini A, Santonico M, Zompanti A, Grasso S, Antonelli Incalzi R, La Grutta S. Repeatability of exhaled breath fingerprint collected by a modern sampling system in asthmatic and healthy children. J Breath Res. 2019 May 1;13(3):036007. doi: 10.1088/1752-7163/ab1765. PMID 30965288